CLINICAL TRIAL: NCT02661919
Title: Assessment of the Emfit Mattress Sensor (L-4060SLC) and Monitor (DVM-GPRS-V2) and Their Acoustic and Cloud Interface Notification Capabilities as a Nocturnal Detection System for Movements Associated With Generalized Tonic-clonic Seizures.
Brief Title: Assessment of the Emfit Mattress Sensor for Detection and Alarm of Night-time Generalized Tonic-clonic Seizures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emfit, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00042423
Record Dates: First submitted 2014-03-14; First posted 2016-01-25 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy; Seizure; Seizures; Mattress monitor; Bed monitor; Bed alarm; Generalized tonic-clonic seizure; GTC
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Emfit mattress sensor (Experimental)
  Interventions: Device: Emfit mattress sensor

INTERVENTIONS:
Device: Emfit mattress sensor — Patients who are being monitored in the Epilepsy Monitoring Unit will have an Emfit mattress sensor placed under their mattress and the effectiveness of the alarm system will be tested.

SUMMARY:
Sudden unexpected death in epilepsy (SUDEP) is the most important epilepsy-related mode of death. The exact mechanism of SUDEP is not known. It is thought that cardiac and respiratory factors are involved. Several ways of preventing SUDEP have been identified. These include seizure control, stress reduction, physical activity, family's ability to perform CPR, and night supervision.

A mattress alarm system that monitors nocturnal seizures can alert family members of night time seizure activity. Thus, a family member could provide aid and therefore potentially avoid SUDEP. The Emfit monitor is intended to perform these tasks.

Investigators tested the Emfit mattress monitor DVM-GPRS-V2 in combination with the Emfit bed sensor L-4060SL in the epilepsy monitoring unit and were able to demonstrate that the device has a high predictive value for detection of generalized convulsions and that it can notify caregivers in the early stages of convulsive activity.

This study will further investigate the upgraded (connected to a cloud server via an integrated cellular GPRS module) Emfit mattress monitor DVM-GPRS-V2 and the upgraded Emfit mattress sensor L-4060SLC in combination with an acoustic and new cloud-based notification system.

ELIGIBILITY:
Inclusion Criteria:

* Overnight Epilepsy Monitoring Unit admission

Exclusion Criteria:

* 12 hours or shorter Epilepsy Monitoring Unit admission

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Alarm effectiveness | 22 months
  Investigators are testing the efficacy of the Emfit mattress monitor acoustic notifications for detecting GTC seizures. During video-eeg monitoring clinically detected GTC seizures are listed. These records are compared to Emfit monitor sound notications detected at video recordings. The true-positive, false-positive and false-negative calculations are primary outcome.

SECONDARY OUTCOMES:
Seizure type distinction | 10 months
  Investigators are testing the Emfit matters sensor acoustic notifications efficacy for detecting other than GTC type seizures (partial seizures, non-epileptic events). Investigators are testing the efficacy of the Emfit mattress monitor acoustic notifications for clinically detected seizures. During video-eeg monitoring clinically detected other than GTC type seizures are listed. These records are compared to Emfit monitor sound notications detected at video recordings. The true-positive, false-positive and false-negative calculations are outcome. False-positive notifications are excluded if patient video recording shows rhytmic movement due patient being awake and performing day-time other activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan U. Schuele, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Narechania AP, Garic II, Sen-Gupta I, Macken MP, Gerard EE, Schuele SU. Assessment of a quasi-piezoelectric mattress monitor as a detection system for generalized convulsions. Epilepsy Behav. 2013 Aug;28(2):172-6. doi: 10.1016/j.yebeh.2013.04.017. Epub 2013 Jun 7. PMID 23747502